CLINICAL TRIAL: NCT04686344
Title: Sonography of the Optic Nerve Sheath Diameter for Comparison Between the Effects of Continuous Infusion of 3%Hypertonic Saline With Intermittent Boluses Versus in Patients With Traumatic Brain Injury.
Brief Title: Point of Care Optic Nerve Sheath Ultrasound to Assess Intracranial Pressure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-383-2020
Record Dates: First submitted 2020-12-19; First posted 2020-12-28 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Optic Nerve Sheath; Hypertonic Saline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic saline continuous infusion Group (Active Comparator): will receive Hypertonic saline continuous infusion
  Interventions: Drug: continuous infusion of Hypertonic saline
- Hypertonic saline intermittent boluses Group (Active Comparator): will receive Hypertonic saline intermittent boluses for 48 hours
  Interventions: Drug: intermittent boluses of Hypertonic saline

INTERVENTIONS:
Drug: intermittent boluses of Hypertonic saline — intermittent boluses every 6 hours over 30 min for 48 hours
  Arms: Hypertonic saline intermittent boluses Group
Drug: continuous infusion of Hypertonic saline — continuous infusion over a period of 48 hours
  Arms: Hypertonic saline continuous infusion Group

SUMMARY:
Elevated intracranial pressure (ICP) is one of the most common symptoms encountered in a variety of traumatic injuries and diseases. Any tissue swelling within the rigid confines of the skull results in increased ICP, which may lead to life-threatening structural alterations in the brain or cerebral blood flow, thus causing oxygen deprivation and ischemia in the brain.

Methods for ICP monitoring can be divided into invasive and noninvasive approaches. In fluid-based systems, external ventricular drainage (EVD) has been considered the gold standard.

Clinicians have found several noninvasive methods that can be used as surrogates for invasive methods for ICP measurement. The optic nerve, as part of the central nervous system, is wrapped by the dural sheath. The optic nerve sheath (ONS) is the continuation of the subarachnoid space at the optic nerve, and its tissues are connected with the subarachnoid space. Thus, an increase in ICP results in a corresponding elevation of the ONS diameter (ONSD).

Hypertonic solutions such as mannitol and hypertonic saline (HTS) are recommended early in the management of ICH after severe TBI . They provide therapeutic benefit along with a wide therapeutic margin. The most recent BTF guidelines stated "although hyperosmolar therapy may lower intracranial pressure, there was insufficient evidence about effects on clinical outcomes to support a specific recommendation, or to support use of any specific hyperosmolar agent".

ELIGIBILITY:
Inclusion Criteria:

1. Patients who having Isolated traumatized brain injury (not for surgical intervention)
2. 3<GCS ≤ 12.
3. Both genders.
4. Age ≥ 18 and ≤ 60Years.
5. Physical status ASA I - III.
6. Cut off value for optic nerve sheath diameter (ONSD) as 5.5 mm to diagnose increase in ICP> 20 mm Hg.

2. Exclusion criteria

1. Patients' first-degree relatives' refusal to sign the consent.
2. GCS (Glasgow coma score) >12 or GCS of 3.
3. Contraindication to hypertonic saline: pregnancy, coagulopathy and cardiac dysfunction.
4. Spinal cord injury, orbital injury, optic nerve injury and optic neuritis.
5. Multi organ affection.
6. Serum Na level ≥ 150 mmol/L at admission to ICU.
7. Hypotension requiring vasopressors to maintain MAP above 60 mmHg.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Diameter of Optic nerve sheath | UP TO 48 HOURS
  assessment tool for Intracranial pressure

SECONDARY OUTCOMES:
intracranial pressure | up to 72 hours
  Rebound increase intracranial pressure
level of Conscious | UP TO 30 DAY
  Glasgow Coma Score : A person's GCS score can range from 3 (completely unresponsive) to 15 (responsive).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo university, Cairo
  - Faculty of Medicine, Cairo University., Cairo

IPD SHARING:
Plan to Share IPD: Undecided